CLINICAL TRIAL: NCT01829282
Title: Implementing Eban II: An Evidence-Based Intervention for HIV Sero-Discordant Couples
Brief Title: Eban II: Intervention for HIV Sero-Discordant Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gail Wyatt, Professor, Dept. of Psychiatry & Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3294930; R01MH093230-01 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Sexually Transmitted Diseases; Disease Transmission, Infectious; Safe Sex; HIV
Keywords: Implementation; HIV; serodiscordant couples; African American; Cultural congruency
MeSH Terms: conditions — Sexually Transmitted Diseases; Communicable Diseases; Safe Sex | interventions — Numbers Needed To Treat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risk Reduction (Experimental): The Risk Reduction group will receive the Eban II Intervention upon enrollment. This group will do the following:
  * Provide HIV and STI test results
  * First Interview
  * Attend 8 sessions - 1 session per week
  * Second interview occurs immediately following the 8th session with HIV and STI tests
  * Third interview occurs 3 months after the 8th session with HIV and STI tests
  Interventions: Behavioral: Risk Reduction
- Waitlist (Active Comparator): The Waitlist group will receive the same intervention after waiting for the Risk Reduction group to complete the entire intervention.
  * Provide HIV and STI test results
  * First Interview
  * No sessions for 8 weeks
  * Second interview and proof of HIV and STI status occurs after the 8 weeks from when you were enrolled
  * Third interview occurs 3 months after the 8th session with HIV and STI tests The Waitlist Group will then be invited to participate in the Risk Reduction group activities.
  * Attend 8 sessions - 1 session per week
  * Fourth interview occurs immediately after the 8th session with HIV and STI tests
  * Fifth interview occurs 3 months after the 8th session with HIV and STI tests
  Interventions: Behavioral: Risk Reduction

INTERVENTIONS:
Behavioral: Risk Reduction

SUMMARY:
This study focuses on the implementation of an evidence-based HIV risk reduction intervention for HIV-serodiscordant, heterosexual African American couples ("Eban II") in two geographic areas (Northern and Southern California - roughly, Alameda and Los Angeles Counties) that have a high prevalence of HIV infection and risk conditions among African Americans.

The Specific Aims are as follows:

1. To evaluate implementation of Eban for HIV serodiscordant African American couples in 10 CBOs in California. To do this, we will document the implementation process and identify barriers and facilitators to Eban's adoption and use by the CBOs. We will interview 200 staff at CBOs to obtain this information.
2. To evaluate the effect of Eban on behavioral and biological outcomes among 180 couples, specifically incidents of protected sex, proportion of condom use, and incident sexually transmitted infections. Eban will be assessed using a randomized delayed enrollment (waitlist) control design to evaluate the impact of treatment on outcomes at posttest and 3-month follow-up (i.e., at these 10 CBOs, Eban will be conducted and offered to couples and evaluated for effectiveness - that is, how well it works in the real world.)
3. To determine the cost-effectiveness of implementation of Eban, based on implementation costs and potential cost savings.

DETAILED DESCRIPTION:
The HIV/AIDS epidemic continues to disproportionately affect African Americans. The rate of HIV among African American men is six times the rate for White men and the rate among African American women is almost 15 times the rate for White women. An estimated 56,300 new HIV cases was reported in 2006, of which 49% were among African Americans and 80% were from heterosexual transmission. Sexually transmitted infections (STIs) also disproportionately affect African Americans, further increasing the risk for HIV transmission. Despite the fact that HIV and STIs are primarily transmitted in the context of relationships, few interventions address HIV risk in couples. Furthermore, few evidence-based HIV prevention interventions have been implemented in community-based organizations (CBOs). Thus, there is a substantial need to strengthen the availability and use of relationship oriented prevention interventions in community-based treatment settings.

This study focuses on the implementation of an evidence-based HIV risk reduction intervention for HIV-serodiscordant, heterosexual African American couples ("Eban II") in two geographic areas (Northern and Southern California - roughly, Alameda and Los Angeles Counties) that have a high prevalence of HIV infection and risk conditions among African Americans.

This study builds upon the multi-site, NIMH-funded "Eban" (a Yoruba term for "fence") trial, which tested this culturally congruent intervention versus a control condition among 535 heterosexual HIV serodiscordant couples in four cities. Couples in the intervention had significantly reduced incidents of unprotected sex and an increased proportion of condom use compared to couples in the control condition. Statistical projections from that study suggest that if Eban participants had not received the intervention, six female and four males would have been infected in one year, and 25 females and 15 males would have become HIV-infected in the next 5 years. Based on these successful outcomes in a controlled trial, it is now appropriate to test the effectiveness of the intervention as delivered in community-based setting. Thus, we propose to conduct a study of implementation - a study of methods to promote the uptake of Eban into community-based organizations (CBOs).

The Specific Aims are as follows:

1. To evaluate implementation of Eban for HIV serodiscordant African American couples in 10 CBOs in California. To do this, we will document the implementation process and identify barriers and facilitators to Eban's adoption and use by the CBOs. We will interview 200 staff at CBOs to obtain this information.
2. To evaluate the effect of Eban on behavioral and biological outcomes among 180 couples, specifically incidents of protected sex, proportion of condom use, and incident sexually transmitted infections. Eban will be assessed using a randomized delayed enrollment (waitlist) control design to evaluate the impact of treatment on outcomes at posttest and 3-month follow-up (i.e., at these 10 CBOs, Eban will be conducted and offered to couples and evaluated for effectiveness - that is, how well it works in the real world.)
3. To determine the cost-effectiveness of implementation of Eban, based on implementation costs and potential cost savings.

So please note, there are essentially two levels to this study -- first to see how well community agencies can implement or take up and execute the intervention (thus, the interviews with staff) - and the second, to see how effective Eban is in real world setting. We know it was highly effective in a controlled study but now we need to test how well it works in the "real" world(thus, the testing of the intervention with 180 couples). While doing this, we will also be examining the cost-effectiveness of the intervention in the "real" world setting.

ELIGIBILITY:
Inclusion Criteria:

* Must be in a relationship with study partner for at least 3 months
* Both partners must be 18 years or older
* At least one partner must identify as African American/Black
* One partner must be HIV positive and one partner must be HIV negative
* Must be a heterosexual couple (one biological female and one biological man)
* Not currently expecting a child and not planning on having children within the year.

Exclusion Criteria:

* Less than 18 years old
* No partner
* Couple is not heterosexual
* Insufficient relationship length/commitment
* No reported incidents of unprotected intercourse in the past 90 days
* Neither partner is African American/Black
* One/both partners unaware of others HIV status
* Couple is not serodiscordant
* One/both partners reported partner violence
* HIV diagnosis received recently (less than 3 months)
* One/both partners participated in a HIV Risk Reduction study within the past 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Safe Sex | within 3 months of completion of the intervention
  Proportion of unprotected acts of sex.

CONTACTS AND LOCATIONS:
Overall Officials: Gail E Wyatt, PhD, Principal Investigator — University of California, Los Angeles; John Williams, MD, Study Director — University of California, Los Angeles; Brian Mittman, PhD, Study Director — VA Office of Research and Development; Alison Hamilton, PhD, Study Director — University of California, Los Angeles; Hector Myers, PhD, Study Director — University of California, Los Angeles
Locations (8):
- United States (8):
  - Tarzana Treatment Centers, Long Beach, California
  - AIDS Project Los Angeles, Los Angeles, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - O.A.S.I.S. Clinic, Los Angeles, California
  - HIV Education & Prevention Project of Alameda County, Oakland, California
  - CAL-PEP, Oakland, California
  - Allen Temple, Oakland, California
  - Women Organized to Respond to Life-Threatening Disease, Oakland, California